CLINICAL TRIAL: NCT00759265
Title: Improving Mobility in Diabetic Patients Through Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-3-031
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2010-07

CONDITIONS: Diabetic Patients With Polyneuropathy
Keywords: Muscle strength; Physical activity; Mobility; Gait analysis
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- resistance training (Experimental): During 24 weeks, the patients of the intervention group will participate in a resistance training program. Two subsequent intervention programmes will be offered. Initially the first 12 week resistance trainings stage will aimed at improving function of lower leg muscles; subsequently a more extended programme affecting total limb musculature (lower- and upper leg) will be provided (also 12 weeks).
  During these trainings period, patients will train 3 times a week; once a plenary training session of 1,5 hour provided by a physical therapist. And 2 trainings sessions of half an hour each, by them selves at home.
  Interventions: Other: resistance training
- control (No Intervention): No intervention was prescribed

INTERVENTIONS:
Other: resistance training — During 24 weeks, the patients of the intervention group will participate in a resistance training program. Two subsequent intervention programmes will be offered. Initially the first 12 week resistance trainings stage will aimed at improving function of lower leg muscles; subsequently a more extended programme affecting total limb musculature (lower- and upper leg) will be provided (also 12 weeks).
  During these trainings period, patients will train 3 times a week; once a plenary training session of 1,5 hour provided by a physical therapist. And 2 trainings sessions of half an hour each, by them selves at home.
  Arms: resistance training

SUMMARY:
Impaired mobility is a major health problem affecting many subjects with diabetes mellitus. It is associated with loss of quality of life and it is a strong predictor for poor health outcomes. Reduced lower extremity muscle function, as a consequence of diabetic polyneuropathy, is a major cause of impaired mobility. We hypothesize that a programme of resistance training will counterbalance the effects of polyneuropathy on muscle wasting, and will improve mobility and associated quality of life.

The objective of this study is to develop a resistance training intervention that improves mobility and quality of life in diabetic patients. It is also our intension to achieve a better understanding of the relation between diabetic neuropathy and muscle weakness, limited mobility and quality of life. Moreover, insight will be gained in optimizing training programmes for neuropathic patients.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients with polyneuropathy:
* valkscore >5;
* diabetic type 2;
* age >50 years

Exclusion Criteria:

* muscular related diseases;
* ischemia;
* amputation (except for toe amputation)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-05; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Mobility | 0 month, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Teunis H IJzerman, MSc, Principal Investigator — Maastricht UMC
Locations (1):
- Academic Hospital Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Melai T, Schaper NC, Ijzerman TH, de Lange TL, Willems PJ, Lima Passos V, Lieverse AG, Meijer K, Savelberg HH. Lower leg muscle strengthening does not redistribute plantar load in diabetic polyneuropathy: a randomised controlled trial. J Foot Ankle Res. 2013 Oct 18;6(1):41. doi: 10.1186/1757-1146-6-41. PMID 24138784